CLINICAL TRIAL: NCT06787924
Title: Effect of Collagen Supplements on Dermal Collagen Content Within Skin Biopsies of Plastic Surgery and Metabolic Bariatric Surgery Patients
Brief Title: Impact of Collagen Supplements on Dermal Collagen in Plastic and Bariatric Surgery Patients
Acronym: COLLAGEN
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: General Committee of Teaching Hospitals and Institutes, Egypt (Other Government)
Responsible Party: Principal Investigator, Mohamed Hany Ashour, Professor, surgeon, General Committee of Teaching Hospitals and Institutes, Egypt
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Collagen_rct_alexandria_hany
Record Dates: First submitted 2025-01-09; First posted 2025-01-22 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Bariatric Surgery; Abdominoplasty; Collagen Synthesis; Skin Physiology; Randomized Controlled Trial; Tissue Remodeling
Keywords: bariatric surgery; collagen supplement; plastic surgery; abdominoplasty; skin; skin quality
MeSH Terms: interventions — Starch

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Starch
  Interventions: Dietary Supplement: Starch
- Collagen (Experimental): Collagen supplement

INTERVENTIONS:
Dietary Supplement: Collagen hydrolyzed peptides — bovine collagen peptides
Dietary Supplement: Starch — Starch placebo
  Arms: Placebo

SUMMARY:
This study aims to evaluate the effects of oral collagen supplementation on dermal collagen content in skin biopsies of patients undergoing abdominoplasty. Using a randomized controlled trial (RCT) design, participants from metabolic bariatric surgery (MBS) and plastic surgery groups will receive either collagen supplements or a placebo for several weeks. Biopsies will be collected pre-intervention and during surgery to compare collagen levels between groups and to baseline. The primary objective is to determine if collagen supplementation significantly enhances dermal collagen deposition compared to placebo and initial levels.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-75 years after metabolic bariatric surgery.
* Patients will be randomly selected from the hospital's electronic patient system.

Exclusion Criteria:

* 1. Allergies or Sensitivities:

  * Patients with known allergies or hypersensitivity to collagen or any components of the collagen supplements (e.g., bovine, marine sources).

    2. Chronic Skin Conditions:
  * Participants with skin disorders that could influence collagen production or degradation (e.g., psoriasis, eczema, scleroderma) should be excluded as these conditions might interfere with the study's outcomes.

    3. Autoimmune or Connective Tissue Diseases:
  * Patients with autoimmune diseases (e.g., lupus, rheumatoid arthritis) or connective tissue disorders (e.g., Ehlers-Danlos syndrome) might exhibit abnormal collagen metabolism and could confound the study's results.

    4. Use of Collagen or Nutritional Supplements:
  * Participants currently taking collagen supplements or other nutritional supplements (e.g., vitamin C, glucosamine, chondroitin) that could affect collagen synthesis or turnover should be excluded. A washout period may be required for those who have recently used such supplements.

    5. Hormonal Treatments or Medications:
  * Patients on treatments that could affect collagen metabolism (e.g., corticosteroids, hormone replacement therapy, anabolic steroids) should be excluded, as these could alter the body's collagen production or degradation.

    6. Pregnancy or Lactation:
  * Pregnant or breastfeeding women should be excluded due to the physiological changes during pregnancy and lactation that could affect collagen metabolism.

    7. Major Surgeries or Trauma:
  * Recent major surgeries or significant trauma within the last 6-12 months, especially those involving connective tissue repair, as these could alter collagen levels independently of supplementation.

    8. Smoking:
  * Smokers or individuals who have recently quit smoking, as smoking is known to reduce collagen synthesis and impair skin healing.

    9. Chronic Illnesses:
  * Patients with chronic illnesses such as diabetes, liver disease, or kidney disease, which could impair collagen metabolism or affect skin health.

    10. Uncontrolled Metabolic Disorders:
  * Participants with uncontrolled metabolic disorders (e.g., severe obesity, untreated hyperlipidemia) may have altered collagen metabolism and should be excluded unless specifically studied.

    11. Participation in Other Clinical Trials:
  * Patients currently enrolled in other clinical trials involving supplements, medications, or procedures that could interfere with the study outcomes should be excluded.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 102 (Estimated)
Dates: Start 2025-04-15 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2025-12-15 (Estimated)

PRIMARY OUTCOMES:
Assessment of Wound Healing Parameters vascularity | Biopsy during surgery
  Wound healing will be evaluated using the single Vancouver Scar Scale (VSS), a validated tool for assessing scar quality. The VSS includes 1. vascularity with higher scores indicating more severe scar formation. This scale will allow for an objective evaluation of the appearance and functional quality of the wound healing in both the collagen supplement and placebo groups. The VSS has been widely used in clinical research for assessing scars in burn patients and offers a standardized approach to scar evaluation
Assessment of Wound Healing Parameters pigmentation | Biopsy during surgery
  Wound healing will be evaluated using the single Vancouver Scar Scale (VSS), a validated tool for assessing scar quality. The VSS includes 2. pigmentation, with higher scores indicating more severe scar formation. This scale will allow for an objective evaluation of the appearance and functional quality of the wound healing in both the collagen supplement and placebo groups. The VSS has been widely used in clinical research for assessing scars in burn patients and offers a standardized approach to scar evaluation
Assessment of Wound Healing Parameters thickness | Biopsy during surgery
  Wound healing will be evaluated using the single Vancouver Scar Scale (VSS), a validated tool for assessing scar quality. The VSS includes 3. thickness, with higher scores indicating more severe scar formation. This scale will allow for an objective evaluation of the appearance and functional quality of the wound healing in both the collagen supplement and placebo groups. The VSS has been widely used in clinical research for assessing scars in burn patients and offers a standardized approach to scar evaluation
Assessment of Wound Healing Parameters pliability | Biopsy during surgery
  Wound healing will be evaluated using the single Vancouver Scar Scale (VSS), a validated tool for assessing scar quality. The VSS includes 4. pliability with higher scores indicating more severe scar formation. This scale will allow for an objective evaluation of the appearance and functional quality of the wound healing in both the collagen supplement and placebo groups. The VSS has been widely used in clinical research for assessing scars in burn patients and offers a standardized approach to scar evaluation

SECONDARY OUTCOMES:
Serum Parameters hydroxyproline | biopsy during surgery
  Total serum hydroxyproline, a marker of collagen degradation and turnover, will be measured in both the collagen supplement and placebo groups using the colorimetric method.
  This well-established technique provides accurate quantification of hydroxyproline levels, which will be used to infer collagen metabolism. Hydroxyproline levels will be compared between the groups using appropriate statistical tests to determine the impact of collagen supplementation on systemic collagen turnover.
  Potential confounding factors, such as dietary gelatin intake and conditions like hepatic fibrosis, which can influence hydroxyproline levels, will be carefully controlled for.
  These factors will be considered exclusion criteria to ensure the reliability of the serum hydroxyproline measurements

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Hany Ashour, professor, MD, Principal Investigator — Alexandria University
Locations (1):
- Facility Name: The surgical department of Medical Research Institute Hospital, Alexandria University, Alexandria, Facility, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The analysis will be performed on a blinded dataset after completing the medical/scientific review. All protocol violations will be identified and resolved, and the dataset will be declared complete. All data will be collected in a data management system (Castor EDC, Amsterdam, The Netherlands; https://www.castoredc.com), handled according to Good Clinical Practice guidelines, Data Protection Directive certificate, and complied with Title 21 CFR Part 11. Furthermore, the data centers where all the research data will be stored are certified according to ISO27001, ISO9001, and Dutch NEN7510
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Available at PI for protocol and SAP ICF, CSR and analytic code after study completion
Access Criteria: Available at PI

REFERENCES:
- [Background] Zague V, de Freitas V, da Costa Rosa M, de Castro GA, Jaeger RG, Machado-Santelli GM. Collagen hydrolysate intake increases skin collagen expression and suppresses matrix metalloproteinase 2 activity. J Med Food. 2011 Jun;14(6):618-24. doi: 10.1089/jmf.2010.0085. Epub 2011 Apr 11. PMID 21480801
- [Background] Sanchez A, Blanco M, Correa B, Perez-Martin RI, Sotelo CG. Effect of Fish Collagen Hydrolysates on Type I Collagen mRNA Levels of Human Dermal Fibroblast Culture. Mar Drugs. 2018 Apr 26;16(5):144. doi: 10.3390/md16050144. PMID 29701725
- [Background] Liu Z, Li Y, Song H, He J, Li G, Zheng Y, Li B. Collagen peptides promote photoaging skin cell repair by activating the TGF-beta/Smad pathway and depressing collagen degradation. Food Funct. 2019 Sep 1;10(9):6121-6134. doi: 10.1039/c9fo00610a. Epub 2019 Sep 9. PMID 31497829
- [Background] Wang X, Hong H, Wu J. Hen collagen hydrolysate alleviates UVA-induced damage in human dermal fibroblasts. Journal of Functional Foods. 2019;63:103574.
- [Background] Mosanya AO, Olasehinde O, Odujoko OO, Etonyeaku AC, Adumah CC, Agbakwuru EA. Comparative study of collagen and elastin content of abdominal wall fascia in inguinal hernia and non-hernia patients in an African population. Hernia. 2020 Dec;24(6):1337-1344. doi: 10.1007/s10029-020-02238-y. Epub 2020 Jun 2. PMID 32488528
- [Background] Aguilar-Toala JE, Hernandez-Mendoza A, Gonzalez-Cordova AF, Vallejo-Cordoba B, Liceaga AM. Potential role of natural bioactive peptides for development of cosmeceutical skin products. Peptides. 2019 Dec;122:170170. doi: 10.1016/j.peptides.2019.170170. Epub 2019 Sep 28. PMID 31574281